CLINICAL TRIAL: NCT01011764
Title: Autism Intervention Research Network on Behavior Health (AIR-B): Study of Peer Relationships at School
Brief Title: Study of Peer Relationships at School
Acronym: HRSAII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Collaborators: Florida State University (Other); Johns Hopkins University (Other); University of Michigan (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor of Psychological Studies in Education and Psychiatry, Health Resources and Services Administration (HRSA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G09-04-021-01A; UA3MC11055 (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Autism
Keywords: social networks; friendships; autism spectrum disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SKILLS group (Active Comparator): The SKILLS intervention targets a specific set of social skills over 8 bi-weekly sessions. The intervention is delivered to a small group of children with autism at school during lunchtime. The content delivered to the group of young children with autism including lessons developed from a manual by Seattle Children's Hospital Research Foundation. Children are given weekly homework assignments to reinforce the topics discussed in the group sessions.
  Interventions: Behavioral: SKILLS vs ENGAGE
- ENGAGE group (Experimental): The ENGAGE intervention targets two social domains, and two learning contexts. The two social domains are peer acceptance and social engagement with peers. The social group will be small and include children with ASD as well as their typical peers. There will be a greater number of typical peers included to model social behaviors and foster friendships. The typical peers will be selected based on results from the friendship survey and teacher nominations. The two learning contexts are direct instruction in a group social skills format during lunchtime and individualized embedded generalization activities in the school day.
  Interventions: Behavioral: SKILLS vs ENGAGE

INTERVENTIONS:
Behavioral: SKILLS vs ENGAGE — The investigators plan to contrast 2 different models for social skills groups. Each model involves 16 45-minute bi-weekly sessions, twice a week with a small group of children with ASD. Details of the 2 intervention models are described below.

SUMMARY:
The goal of this study is to compare the effects of two separate, manualized group interventions designed to improve social outcomes for young children with autism. The first type of group intervention utilizes a social skill curriculum delivered to a small group of children with autism at their school. This type of group will be referred to as the Skills group (SKILLS intervention). The other intervention delivers a social engagement curriculum at the children's school site and includes children with autism and typically developing peers, from the same school. This type of group will be referred to as the School Engagement Group (ENGAGE intervention).

DETAILED DESCRIPTION:
Once families have decided to join the study, and have completed the informed consent process using the "Social Skills Club - Parent Consent", and once we obtain letters of agreement from participating elementary schools, children with ASD will be randomly assigned to one of two intervention conditions, SKILLS or ENGAGE, led by two trained doctoral students. Since children will be randomized to either the SKILLS or the ENGAGE group, we are hoping to determine the active ingredients for successfully integrating children with autism. For both the SKILLS and the ENGAGE groups, all interventions and observations of children will take place in the target child's school. Thus, upon admission to the project, research personnel will attend the participant's classroom at school, and distribute consent forms titled "Peer Relationships at School - Classroom Parent Consent" to all children in the class. The consenting process should be no more than ten minutes. For those children that return informed consent from their parents, as well as offer assent on the "Children's Classroom Assent" to join to the project, social network measures (including brief demographic information), as well as friendship surveys (Friendships Qualities Scale; FQS), and an emotion measure (loneliness questionnaire) will be distributed at pre-intervention (baseline), post-intervention, and follow-up time points. These measures will take approximately 30-40 minutes per each time point. Graduate students will administer the measures and will make every effort to do so at a convenient time for the teacher and for the classroom to avoid utilizing instructional time. In addition, the efficacy of the treatment interventions will be assessed with ongoing direct behavioral observations at entry, twice during treatment, at exit, and at the 2-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Children are between the ages of 7 and 12 years in grades 2-5.
* Children have a clinical diagnosis of autism or PDD-NOS, and/or meet criteria on the ADOS for ASD or autism.
* Children have an IQ of 70 or above
* Children are fully included in a typical classroom for 80% or more of the school day
* Children are expected to stay in the school or the classroom for the duration of the study.
* Families with low SES and/or from racial/ethnic minority backgrounds

Exclusion Criteria:

* Children must not have additional diagnoses or sensory or motor impairments.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The Friendship Survey | Before treatment, after treatment, and 2 months after treatment

SECONDARY OUTCOMES:
Friendship Qualities Scale | Before treatment, after treatment, and 2 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Connie Kasari, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (5):
- United States (5):
  - University of California, Los Angeles, Los Angeles, California
  - Florida State University, Tallahassee, Florida
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Bauminger N, Kasari C. Loneliness and friendship in high-functioning children with autism. Child Dev. 2000 Mar-Apr;71(2):447-56. doi: 10.1111/1467-8624.00156. PMID 10834476
- [Background] Chamberlain B, Kasari C, Rotheram-Fuller E. Involvement or isolation? The social networks of children with autism in regular classrooms. J Autism Dev Disord. 2007 Feb;37(2):230-42. doi: 10.1007/s10803-006-0164-4. PMID 16855874
- [Background] Kasari C, Freeman SF, Bauminger N, Alkin MC. Parental perspectives on inclusion: effects of autism and Down syndrome. J Autism Dev Disord. 1999 Aug;29(4):297-305. doi: 10.1023/a:1022159302571. PMID 10478729
- [Background] Robertson K, Chamberlain B, Kasari C. General education teachers' relationships with included students with autism. J Autism Dev Disord. 2003 Apr;33(2):123-30. doi: 10.1023/a:1022979108096. PMID 12757351